CLINICAL TRIAL: NCT05525338
Title: Standard Dosed Alectinib Versus Therapeutic Drug Monitoring Guided Alectinib Dosing
Brief Title: Comparison of Standard Dose Alectinib to Alectinib in Adjusted Dose Based on Alectinib Bloodlevels
Acronym: ADAPT ALEC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Amsterdam University Medical Center (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Radboud University Medical Center (Other); The Netherlands Cancer Institute (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202000251; 2020-001737-13 (EudraCT Number); NL9411 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2022-08-26; First posted 2022-09-01 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Drug Monitoring; Carcinoma, Non-Small-Cell Lung; Lung Cancer; Anaplastic Lymphoma Kinase Gene Mutation; Anaplastic Lymphoma Kinase Gene Translocation
Keywords: Alectinib; Randomized Controlled Trial
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — alectinib

STUDY DESIGN:
Intervention Model Description: Both study-arms will receive oral alectinib (Alecensa®, Roche). In arm A (TDM arm), the alectinib dose will be increased if Cmin <435 ng/mL and manageable toxicity. In both arms, alectinib dose can be reduced based on toxicity.
Masking Description: The alectinib Cmin for patients treated in arm B (standard dose arm) will be blinded to participants and care providers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDM-guided dosing arm (Experimental)
  Interventions: Drug: Alectinib
- Standard dose arm (No Intervention): Alectinib plasmaconcentration will be blinded untill the end of the trial. No intervention based on the alectinib plasmaconcentrion will be performed. In case of unacceptable toxicity (i.e. unbearable or persistent grade 2 toxicity and grade 3/4 toxicity), the alectinib dose can be reduced by 150mg BID.

INTERVENTIONS:
Drug: Alectinib — In case of an alectinib plasmaconcentration Cmin <435 ng/mL, determined by TDM, and manageable toxicity, the alectinib dose will be increased with 150mg BID up to a maximum of 900mg BID. In case of unacceptable toxicity (i.e. unbearable or persistent grade 2 toxicity and grade 3/4 toxicity), the alectinib dose can be reduced by 150mg BID.
  Arms: TDM-guided dosing arm

SUMMARY:
The ADAPT ALEC randomized controlled trial (RCT) is performed in patients with Anaplastic Lymphoma Kinase (ALK) positive non-small cell lung cancer (NSCLC). The RCT will compare the use of Therapeutic Drug Monitoring (TDM) and dose increases if alectinib 35 ng/Ml (arm A) with standard of care (arm B).

DETAILED DESCRIPTION:
The ADAPT ALEC trial is a phase IV, RCT in patients with ALK positive NSCLC treated with alectinib. A longer median progression free survival (mPFS) is expected in patients treated with standard dose alectinib when minimum plasma concentrations (Cmin) of alectinib exceed 435 ng/mL. The ADAPT ALEC trial will investigate whether using therapeutic drug monitoring (TDM) and increasing the dose of alectinib in patients with Cmin <435 ng/mL, will raise the mPFS. We will compare mPFS in the subgroup of patients with an alectinib Cmin <435 ng/mL using TDM and dose increases (arm A) to fixed dosing/standard of care (arm B).

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic NSCLC (stage IIIB to stage IV by AJCC 8th)
* ECOG performance status 0-4
* Histologically or cytology confirmed NSCLC
* Documented ALK rearrangement based on an EMA approved test
* Patients can either be chemotherapy-naïve or have received one line of platinum-based chemotherapy
* Patients with brain or leptomeningeal metastases are allowed on the study if the lesions are asymptomatic without neurological signs and clinically stable for at least 2 weeks without steroid treatment. Patients who do not meet these criteria are not eligible for the study
* Measurable disease (by RECIST criteria version 1.1) prior to the first dose of study treatment
* Signed writte Institutional Review Board (IRB)/Ethical Committee (EC) approved informed consent form, prior to performing any study-related procedures
* Observational other studies are allwoed for patients included in this study
* Local radiotherapy is allowed for pain

Exclusion Criteria:

* Any significant concomitant disease determined by the investigator to be potentially aggravated by the investigational drug
* Consumption of agents which modulate CYP3A4 or agents with potential QT prolonging effects within 14 days prior to admission and during the study (see concomitant medication restrictions)
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study, or absorption of oral medications, or that would, in the opinion of the Principal Investigator, pose an unacceptable risk to the subject in this study.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the patient before trial entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Median progression free survival (mPFS) | mPFS will be assessed through study completion, after 12 months of follow-up.
  PFS is measured from start of treatment to progressive disease, death or lost to follow-up.Patients who did not die or progress, or lost to follow-up, will be censored at their last available date.

SECONDARY OUTCOMES:
Succesfull Therapeutic Drug monitoring | 4 to 6 weeks after dose adjustment based on TDM
  The percentage of succesfull TDM interventions, in which successful is defines as tartget attainment and manageable toxicity.
Overall response rate (ORR) | Response will be assessed every 2-3 months. ORR will be determined after total study completion and 12 months of follow-up
  ORR is the percentage of patients with partial response or complete response, according to RECIST v1.1, of the total treated population.
Median overall survival | Through total study completion, after 12 months of follow-up
  mOS is defined as time from randomization to death from any cause in the total population.
Intracranial PFS | Progressive disease will be assessed once every 2-3 months. Intracranial PFS will be assessed through total study completion, after 12 months of follow-up
  PFS is measured from start of treatment to progressive disease in the brain, death or lost to follow-up. Patients who did not die or progress, or lost to follow-up, will be censored at their last available date.
Patient adherence to alectinib treatment | Through study completion, an average of 2 years
  This will be estimated by pill counts of returned medication as well as a patient diary on drug intake.
Number of adverse events (AE) related to plasma concentration and dose increases | Through total study completion, after 12 months of follow-up
  AE's will be defined using CTCAE v5.0. Number of AE's in the subgroups of patients with Cmin <435 ng/mL compared to Cmin >= 435 ng/ML, and in patients who did and who did not receive a TDM-guided dose increase.
European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC QLQ-C30) and the the Quality of Life Questionnaire-Lung Cancer 13 (EORTC QLQ-LC-13) module | Questionnaires will be filled in at baseline and every 3 months thereafter through study completion, an average of 2 years.
  Mean change from baseline in EORTC QLQ-C30 and QLQ-LC13 scores
European Quality of Life Five Dimensions with five levels (EQ-5D-5L) questionnaire | Questionnaire will be filled in at baseline and every 3 months thereafter through study completion, an average of 2 years.
  Mean change from baseline in EQ-5D-5L score
Incremental cost-effectiveness ratio (ICER) | Through total study completion, after 12 months of follow-up
  The ICER is the final outcome of the comparative cost-effectiveness analysis performed using a health-state transition model to compare costs and effectiveness between both study arms.
Alectinib M4 protein | Through total study completion, after 12 months of follow-up
  Alectinib M4 plasmaconcentrations in relation to alectinib plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: A.J. van der Wekken, PhD, Principal Investigator — University Medical Center Groningen
Locations (8):
- Gustave Roussy, Villejuif, Val-de-Marne, France
- Netherlands (7):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht University Medical Center +, Maastricht, Limburg
  - The Netherlands Cancer Institute, Amsterdam, North Holland
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will only be shared upon reasonable request from the Principal Investigator at the UMCG, who will discuss the request with the ADAPT ALEC study team.
Supporting Information: Study Protocol
Time Frame: The study protocol will be available after ending of the study and publication of the manuscript ending 5 years after article publication.
Access Criteria: For individual participant data meta-analysis

REFERENCES:
- [Derived] Meertens M, Muntinghe-Wagenaar MB, Sikkema BJ, Lopez-Yurda M, Retel VP, Paats MS, Ter Heine R, Schuuring E, Timens W, Touw DJ, van Boven JFM, de Langen AJ, Hashemi SMS, Hendriks LEL, Croes S, van den Heuvel MM, Dingemans AC, Mathijssen RHJ, Smit EF, Huitema ADR, Steeghs N, van der Wekken AJ. Therapeutic drug monitoring guided dosing versus standard dosing of alectinib in advanced ALK positive non-small cell lung cancer patients: Study protocol for an international, multicenter phase IV randomized controlled trial (ADAPT ALEC). Front Oncol. 2023 Mar 9;13:1136221. doi: 10.3389/fonc.2023.1136221. eCollection 2023. PMID 36969063